CLINICAL TRIAL: NCT03692364
Title: Randomized Evaluation of Metal-on-conventional-polyethylene vs Ceramic-on-ceramic Articulating Surfaces in Uncemented Total Hip Arthroplasty: A Radiostereometry Study Including 104 Patients
Brief Title: Evaluation of Metal-on-conventional-polyethylene vs Ceramic-on-ceramic Articulating Surfaces in Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Principal Investigator, Per-Erik Johanson, Researcher, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protesteam_ceram
Record Dates: First submitted 2018-08-20; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Arthroplasty Complications
Keywords: biomaterials; Implant wear; hip arthroplasty; osteolysis; aseptic loosening
MeSH Terms: conditions — Osteolysis

STUDY DESIGN:
Intervention Model Description: Prospective randomized study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Metal-on-conventional polyethylene (Active Comparator): Uncemented hip arthroplasty (ABG-2, Stryker, Mahwah NJ, US) with a CoCr prosthetic femoral head and an acetabular liner made of intermedially cross-linked polyethylene polyethylene (Duration, Stryker, Mahwah, NJ, US).
  Interventions: Device: Metal-on-polyethylene uncemented total hip arthroplasty
- Ceramic-on-ceramic (Experimental): Uncemented hip arthroplasty (ABG-2, Stryker, Mahwah NJ, US) with a prosthetic femoral head and an acetabular liner made of alumina ceramic (Biolox Forte, Ceramtec, Plochingen, Germany).
  Interventions: Device: Ceramic-on-ceramic uncemented hip arthroplasty

INTERVENTIONS:
Device: Ceramic-on-ceramic uncemented hip arthroplasty
  Arms: Ceramic-on-ceramic
Device: Metal-on-polyethylene uncemented total hip arthroplasty
  Arms: Metal-on-conventional polyethylene

SUMMARY:
Polyethylene wear debris from metal-on-polyethylene articulations are one of the main causes of periprosthetic bone loss and non-infectious loosening in total hip arthroplasty. Ceramic articulations have a very low wear rate when measured in the laboratory and the investigator's hypothesis is that hip arthroplasty with an all ceramic articulation will have less osteolysis and wear in addition to equally good fixation and clinical outcome compared to the same hip arthroplasty design with a metal-on-polyethylene joint.

ELIGIBILITY:
Inclusion Criteria:

* primary osteoarthritis
* secondary osteoarthritis caused by idiopathic osteonecrosis, dysplasia or childhood disease (Mb Perthes, epiphysiolysis)

Exclusion Criteria:

* inflammatory arthritis
* hip joint infection

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2003-10-02 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Osteolysis frequency change between 7 and 15 years | Change between 7 to 15 years after surgery
  Osteolysis frequency (%) measured with computed tomography,
Osteolysis size change between 7 and 15 years | Change between 7 and 15 years after surgery
  Osteolysis size (cm3) measured with computed tomography

SECONDARY OUTCOMES:
Articulation wear at 7 years | At 7 years after surgery
  Articulation wear as measured with radiostereometry, mm/year
Articulation wear at 15 years | 15 years after surgery
  Articulation wear as measured with radiostereometry, mm/year
Implant fixation at 7 years | 7 years after surgery
  Stem and cup translation (mm/year) and rotation (degrees/year) measured with radiostereometry
Implant fixation at 15 years | At 15 years after surgery
  Stem and cup translation (mm/year) and rotation (degrees/year) measured with radiostereometry
Clinical function at 7 years | 7 years after surgery
  Harris Hip Score (0-100)
Clinical function at 15 years | 15 years after surgery
  Harris Hip Score (0-100)

IPD SHARING:
Plan to Share IPD: No